CLINICAL TRIAL: NCT06154408
Title: Evaluating the Impact of Omega-3 Fatty Acid Supplementation (Soloways™) on Lipid Profiles in Adults With PPARG Polymorphisms: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Evaluating the Impact of Omega-3 Fatty Acid Supplementation (Soloways™) on Lipid Profiles in Adults With PPARG Polymorphisms
Acronym: SOLIPARG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Center of New Medical Technologies (Other); Triangel Scientific (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SW001
Record Dates: First submitted 2023-11-22; First posted 2023-12-04 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: LDL Hyperlipoproteinemia; Low-Density-Lipoprotein-Type [LDL] Hyperlipoproteinemia; Triglyceride Storage Type I or II Disease
Keywords: PPARG polymorphisms; omega-3 fatty acids; LDL-C; triglycerides; cardiovascular health; personalized medicine
MeSH Terms: interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- omega-3 fatty acids group (Experimental)
  Interventions: Dietary Supplement: omega-3 fatty acids
- placebo group (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: omega-3 fatty acids — The active treatment, supplied by Soloways, LLC., contained omega-3 fatty acids (1000 mg of fish oil, of which 600 mg were eicosapentaenoic acid and 300 mg docosahexaenoic acid) per capsule. The subjects will take 2 capsules daily.
  Other Names: omega-3 fatty acids 1000mg
  Arms: omega-3 fatty acids group
Dietary Supplement: Placebo — placebo capsules identical in appearance, matched for color coating, shape, and size with omega-3 fatty acids capsule
  Arms: placebo group

SUMMARY:
In this study, 102 patients will be evenly randomized into two groups: one set to receive omega-3 fatty acids and the other a placebo. The process will be blinded, ensuring that neither the researchers nor the participants will know which group they are in. Each participant will take two capsules daily for a duration of 90 days, with the active group receiving capsules containing 1000 mg of fish oil each. All participants will be instructed to maintain their usual diet, lifestyle, and medication regimen.

At the beginning and end of the study, various health assessments, including lipid panels and C-reactive protein measurements, will be conducted. Additionally, DNA samples will be collected for genotyping to identify patients with specific PPARG gene polymorphisms, leading to the creation of four distinct subgroups: those receiving omega-3 with and without polymorphisms, and those receiving placebo with and without polymorphisms.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 75;
* ( LDL-C level between 70 and 190 mg/dL, confirmed in at least two sequential checks conducted within the last six months prior to signing the consent form.

Exclusion Criteria:

* Personal history of cardiovascular disease or hight risk (≥ 20%);
* Triglycerides (TG) ≥ 400 mg/dL;
* Obesity (Body Mass Index > 32 kg/m2);
* Assumption of lipid-lowering drugs or supplements affecting lipid metabolism within the last three months;
* Diabetes mellitus;
* Known severe or uncontrolled thyroid, liver, renal, or muscle diseases.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
the percent change in LDL-C for omega-3 fatty acids among patients with PPARG polymorphism | 90 days
  the percent change in LDL-C for omega-3 fatty acids compared with placebo among patients with PPARG polymorphism

SECONDARY OUTCOMES:
the percent change in hsCRP | 90 days
  the percent change in hsCRP for omega-3 fatty acids compared with placebo among patients with PPARG polymorphism
the percent change in High-density lipoprotein cholesterol | 90 days
  the percent change in High-density lipoprotein cholesterol for omega-3 fatty acids compared with placebo among patients with PPARG polymorphism
the percent change in total cholesterol the percent change in total cholesterol | 90 days
  the percent change in total cholesterol for omega-3 fatty acids compared with placebo among patients with PPARG polymorphism
the percent change in serum triglycerides | 90 days
  the percent change in serum triglycerides for omega-3 fatty acids compared with placebo among patients with PPARG polymorphism

CONTACTS AND LOCATIONS:
Locations (1):
- Center of New Medical Technologies, Novosibirsk, Novosibisk Region, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pokushalov E, Ponomarenko A, Bayramova S, Garcia C, Pak I, Shrainer E, Voronina E, Sokolova E, Johnson M, Miller R. Evaluating the Impact of Omega-3 Fatty Acid (SolowaysTM) Supplementation on Lipid Profiles in Adults with PPARG Polymorphisms: A Randomized, Double-Blind, Placebo-Controlled Trial. Nutrients. 2023 Dec 27;16(1):97. doi: 10.3390/nu16010097. PMID 38201926
- See also: DOI: 10.3390/nu16010097 — http://pubmed.ncbi.nlm.nih.gov/38201926/